CLINICAL TRIAL: NCT06295614
Title: Study on Preliminary Safety and Efficacy of the ARC-IM Therapy to Alleviate Locomotor Deficits in People With Parkinson's Disease
Acronym: SPARKL
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ecole Polytechnique Fédérale de Lausanne (Other)
Responsible Party: Principal Investigator, Jocelyne Bloch, Prof., Centre Hospitalier Universitaire Vaudois
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SPARKL
Record Dates: First submitted 2024-02-20; First posted 2024-03-06 (Actual); Last update posted 2025-07-11 (Actual); Status verified 2025-07

CONDITIONS: Parkinson Disease
Keywords: Parkinson Disease; Spinal Cord Stimulation; Epidural Spinal Stimulation
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Intervention Model Description: Single-site, single-arm, non-blinded, non-randomized, interventional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- All participants (Experimental): All participants enrolled in the study will receive the same intervention.
  The first year of the study consists of the following phases: enrolment, baseline assessments, surgical implantation of the ARC-IM stimulation device, configuration sessions for stimulation, in-clinic and at-home rehabilitation, and a home-use phase. It is followed by 3 years of safety follow-up.
  Assessments will be planned throughout the course of the study and at baseline, the end of the optimization phase, the end of the rehabilitation phase, and after 12 months post-surgery.
  Interventions: Device: ARC-IM System implantation

INTERVENTIONS:
Device: ARC-IM System implantation — Implantation of a stimulation lead on the lumbar level of the spinal cord and implantation of a neurostimulator in the abdominal region.

SUMMARY:
The purpose of this clinical trial is to assess the preliminary safety and efficacy of the ARC-IM spinal cord stimulation therapy in alleviating locomotor deficits in individuals with Parkinson's disease. The ARC-IM Therapy employs epidural electrical stimulation (EES) to modulate leg muscle recruitment, with the aim of improving mobility deficits. The ultimate goal is to enhance the quality of life of people with Parkinson's disease.

DETAILED DESCRIPTION:
The progression of Parkinson's Disease (PD) is often marked by the development of severe locomotor deficits, including gait impairments, which significantly affect patients' independence and are not effectively addressed by current treatments. The STIMO-PARKINSON (NCT04956770) clinical trial has shown promising results with epidural electrical stimulation (EES) in significantly reducing these locomotor deficits in Parkinson's Disease patients.

Building on these findings, the SPARKL clinical study aims to further this research. The SPARKL study aims to enroll six individuals with advanced Parkinson's Disease to assess the safety and efficacy of the novel ARC-IM Therapy. This new therapy has been designed to overcome previous technological limitations and facilitate its home-use.

This study will take place at the Lausanne University Hospital (CHUV, Switzerland). The total duration of the study is 4 years per participant. The study intervention consists of several phases preceded by pre-screening. The first year involves an intensive participation, consisting of the following phases: enrolment and baseline, surgical implantation of the stimulation device, a main study phase that includes stimulation configuration sessions and both in-clinic and at-home rehabilitation, and finally the home-use phase. This will be succeeded by 3 years of safety follow-up, during which the participant can use the stimulation device in their daily life, subject to investigator approval.

Throughout the study, the investigators will conduct assessments at various stages of each participant's journey in the study. These assessments will be used to assess the preliminary safety and efficacy of the ARC-IM therapy at alleviating locomotor deficits.

ELIGIBILITY:
Inclusion Criteria:

* Typical form of Parkinson's Disease with II-IV Hoehn-Yahr stage with standard therapy,
* Suffering from debilitating locomotor deficits, including gait impairments of either postural instability and/or freezing of gait, despite optimal medical management,
* 18 years of age or older,
* Able to understand and interact with the study team in French or English,
* Must use safe contraception for women of childbearing capacity,
* Must agree to comply in good faith with all conditions of the study and to attend all required study trainings and visits.
* Must provide and sign the study's Informed Consent prior to any study-related procedures.

Exclusion Criteria:

* Atypical forms of Parkinson's Disease (such as Multiple System Atrophy or Progressive Supranuclear Palsy),
* Secondary causes of gait problems independent of Parkinson's Disease,
* Inability to follow study procedures,
* Unstable or significant medical condition that is likely to interfere with study procedures or likely to confound study endpoint evaluations as determined by the Investigator,
* History of major psychiatric disorders or major neurocognitive disorder as considered by the Investigators in accordance with treating physician and treating neurologist,
* Major change in PD treatment planned until the end of the main study phase (such as Deep Brain Stimulation or dopamine-pump implantation),
* Diseases and conditions that would increase the morbidity and mortality of the implantation surgery,
* Spinal anatomical abnormalities precluding surgery,
* History of drug or alcohol abuse in the past 5 years,
* Life expectancy of less than 12 months,
* Pregnant or breast feeding,
* Intention to get pregnant during the course of the study,
* Indication requiring frequent Magnetic Resonance Imaging (MRI),
* Experimental treatment taken in the past 5 years,
* Participation in another interventional study,
* Enrolment of the investigator, his/her family members, employees, and other dependent persons.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Estimated)
Dates: Start 2024-02-14 (Actual); Primary Completion 2029-04-01 (Estimated); Study Completion 2029-04-01 (Estimated)

PRIMARY OUTCOMES:
Occurrence of serious adverse events and adverse events that are deemed related or possibly related to the study procedures or to the investigational system. | From enrollment until end of safety follow-up phase (4 years)
  Assess the safety of the ARC-IM Therapy at alleviating locomotor deficits in people with Parkinson's Disease.

SECONDARY OUTCOMES:
10-meter walk test | Baseline (before surgery), Short-Term assessments (~1 month post-surgery) and Follow-Up assessments (~4 & 11 months post-surgery)
  To assess gait speed. Measurement tool: time (s)
6-minute walk test | Baseline (before surgery), Short-Term assessments (~1 month post-surgery) and Follow-Up assessments (~4 & 11 months post-surgery)
  To assess endurance. Measurement tool: distance (m)
Timed up and Go and its cognitive version | Baseline (before surgery), Short-Term assessments (~1 month post-surgery) and Follow-Up assessments (~4 & 11 months post-surgery)
  To assess freezing of gait prevalence. Measurement tool: time (s)
Freezing of gait circuit | Baseline (before surgery), Short-Term assessments (~1 month post-surgery) and Follow-Up assessments (~4 & 11 months post-surgery)
  To assess freezing of gait prevalence. Measurement tool: time (s)
Kinematic analysis | Baseline (before surgery), Short-Term assessments (~1 month post-surgery) and Follow-Up assessments (~4 & 11 months post-surgery)
  Gait circuit to assess gait kinematic. Measurement tool: changes in position and orientation of the body through sensors (mm)
Muscle analysis | Baseline (before surgery), Short-Term assessments (~1 month post-surgery) and Follow-Up assessments (~4 & 11 months post-surgery)
  Gait circuit to assess muscle activity. Measurement tool: muscle activity through sensors (mV)
Mini Balance Evaluation Systems Test (mini-BESTest) | Baseline (before surgery), Short-Term assessments (~1 month post-surgery) and Follow-Up assessments (~4 & 11 months post-surgery)
  4-item test to assess balance. Measurement tool: total score
Movement Disorders Society Unified Parkinson's Disease Rating Scale (MDS-UPDRS) Part III | Baseline (before surgery), Short-Term assessments (~1 month post-surgery) and Follow-Up assessments (~4 & 11 months post-surgery)
  19 item-test to assess the course of Parkinson's Disease. Measurement tool: total score from 0 up to 132. Low score means a better outcome.
King's Parkinson's disease Pain Scale (KPPS) | Baseline (before surgery), Short-Term assessments (~1 month post-surgery) and Follow-Up assessments (~4 & 11 months post-surgery)
  7-item questionnaire to assess daily life performance. Measurement tool: total score 0 up to 168. Low score means a better outcome.
The Movement Disorders Society Unified Parkinson's Disease Rating Scale (MDS-UPDRS) Part IA & IV Part I, II & IV. | Baseline (before surgery), Short-Term assessments (~1 month post-surgery) and Follow-Up assessments (~4 & 11 months post-surgery)
  3-part questionnaire to assess daily life performance. Measurement tool: total score from 0 up to 128. Low score means a better outcome.
Parkinson's Disease Questionnaire-39 (PDQ-39) | Monthly, from the start of the study until the end of the home-use phase (~12 months)
  39-item questionnaire to assess daily life performance. Measurement tool: total score from 0 up to 100. Low score means a better outcome.
Activities specific Balance Confidence Questionnaire (ABC-Q) | Monthly, from the start of the study until the end of the home-use phase (~12 months)
  16-item questionnaire to assess daily life performance. Measurement tool: total score from 0 up to 100. High score means a better outcome.
The Freezing of Gait Questionnaire (FOG-Q) | Monthly, from the start of the study until the end of the home-use phase (~12 months)
  6-item questionnaire to assess daily life performance. Measurement tool: total score 0 up to 24. High score means a better outcome.
Home-use kinematic monitoring | Weekly, from the start of the study until the end of the home-use phase (~12 months)
  To assess gait pattern in ecological environment. Measurement tool: changes in position and orientation of the feet through sensors placed on shoes (mm)
Daily falls tracking | Weekly, from the start of the study until the end of the home-use phase (~12 months)
  To assess daily falls. Measurement tool: number of falls
Satisfaction questionnaire | Monthly, from the Short-Term assessments (~1 month post-surgery) until the end of the home-use phase (~12 months)
  16-item questionnaire to collect feedback from the therapy. Measurement tool: total score from 0 up to 100.
User Evaluation of Satisfaction with technology (QUEST 2.0) | Follow-Up assessments (~4 & 11 months post-surgery)
  12-item questionnaire to assess usability of the therapy. Measurement tool: total score from 12 up to 60. Low score means a better outcome.
System Usability Scale (SUS) | Follow-Up assessments (~4 & 11 months post-surgery)
  Questionnaire to assess usability of the therapy. Measurement tool: total score from 0 to 100. High score means a better outcome.

OTHER OUTCOMES:
Nerve conduction studies (NCS) | Baseline assessments
  To assess status of peripheral nervous system. Measurement tool: electrical activity in the nerve (mV)
Somato-sensory evoked potential (SSEP) | Short-term assessments (~1 month post-surgery)
  To assess the transmission of electrical activity from a touch stimulation. Measurement tool: electrical activity in the nerve (mV)
Cortical signal recording | After surgery, until 18 weeks post-surgery
  To assess changes in brain activity patterns. Measurement tool: electrical activity in the brain (mV)
Kinematic analysis in different therapeutic conditions | After surgery, until 18 weeks post-surgery
  Gait circuit to assess gait kinematic changes. Measurement tool: changes in position and orientation of the body through sensors (mm)
Muscle analysis in different therapeutic conditions | After surgery, until 18 weeks post-surgery
  Gait circuit to assess muscle activity change. Measurement tool: muscle activity through sensors (mV)

CONTACTS AND LOCATIONS:
Overall Officials: Jocelyne Bloch, MD, Principal Investigator — Centre hospitalier universitaire vaudois (CHUV)
Locations (1):
- Centre Hospitalier Universitaire Vaudois (CHUV), Lausanne, Canton of Vaud, Switzerland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Yakovenko S, Mushahwar V, VanderHorst V, Holstege G, Prochazka A. Spatiotemporal activation of lumbosacral motoneurons in the locomotor step cycle. J Neurophysiol. 2002 Mar;87(3):1542-53. doi: 10.1152/jn.00479.2001. PMID 11877525
- [Background] Bloem BR, Hausdorff JM, Visser JE, Giladi N. Falls and freezing of gait in Parkinson's disease: a review of two interconnected, episodic phenomena. Mov Disord. 2004 Aug;19(8):871-84. doi: 10.1002/mds.20115. PMID 15300651
- [Background] Schaafsma JD, Giladi N, Balash Y, Bartels AL, Gurevich T, Hausdorff JM. Gait dynamics in Parkinson's disease: relationship to Parkinsonian features, falls and response to levodopa. J Neurol Sci. 2003 Aug 15;212(1-2):47-53. doi: 10.1016/s0022-510x(03)00104-7. PMID 12809998
- [Background] Rowald A, Komi S, Demesmaeker R, Baaklini E, Hernandez-Charpak SD, Paoles E, Montanaro H, Cassara A, Becce F, Lloyd B, Newton T, Ravier J, Kinany N, D'Ercole M, Paley A, Hankov N, Varescon C, McCracken L, Vat M, Caban M, Watrin A, Jacquet C, Bole-Feysot L, Harte C, Lorach H, Galvez A, Tschopp M, Herrmann N, Wacker M, Geernaert L, Fodor I, Radevich V, Van Den Keybus K, Eberle G, Pralong E, Roulet M, Ledoux JB, Fornari E, Mandija S, Mattera L, Martuzzi R, Nazarian B, Benkler S, Callegari S, Greiner N, Fuhrer B, Froeling M, Buse N, Denison T, Buschman R, Wende C, Ganty D, Bakker J, Delattre V, Lambert H, Minassian K, van den Berg CAT, Kavounoudias A, Micera S, Van De Ville D, Barraud Q, Kurt E, Kuster N, Neufeld E, Capogrosso M, Asboth L, Wagner FB, Bloch J, Courtine G. Activity-dependent spinal cord neuromodulation rapidly restores trunk and leg motor functions after complete paralysis. Nat Med. 2022 Feb;28(2):260-271. doi: 10.1038/s41591-021-01663-5. Epub 2022 Feb 7. PMID 35132264
- [Background] Wagner FB, Mignardot JB, Le Goff-Mignardot CG, Demesmaeker R, Komi S, Capogrosso M, Rowald A, Seanez I, Caban M, Pirondini E, Vat M, McCracken LA, Heimgartner R, Fodor I, Watrin A, Seguin P, Paoles E, Van Den Keybus K, Eberle G, Schurch B, Pralong E, Becce F, Prior J, Buse N, Buschman R, Neufeld E, Kuster N, Carda S, von Zitzewitz J, Delattre V, Denison T, Lambert H, Minassian K, Bloch J, Courtine G. Targeted neurotechnology restores walking in humans with spinal cord injury. Nature. 2018 Nov;563(7729):65-71. doi: 10.1038/s41586-018-0649-2. Epub 2018 Oct 31. PMID 30382197
- [Background] Capogrosso M, Wenger N, Raspopovic S, Musienko P, Beauparlant J, Bassi Luciani L, Courtine G, Micera S. A computational model for epidural electrical stimulation of spinal sensorimotor circuits. J Neurosci. 2013 Dec 4;33(49):19326-40. doi: 10.1523/JNEUROSCI.1688-13.2013. PMID 24305828
- [Background] Moraud EM, Capogrosso M, Formento E, Wenger N, DiGiovanna J, Courtine G, Micera S. Mechanisms Underlying the Neuromodulation of Spinal Circuits for Correcting Gait and Balance Deficits after Spinal Cord Injury. Neuron. 2016 Feb 17;89(4):814-28. doi: 10.1016/j.neuron.2016.01.009. Epub 2016 Feb 4. PMID 26853304
- [Background] Capogrosso M, Wagner FB, Gandar J, Moraud EM, Wenger N, Milekovic T, Shkorbatova P, Pavlova N, Musienko P, Bezard E, Bloch J, Courtine G. Configuration of electrical spinal cord stimulation through real-time processing of gait kinematics. Nat Protoc. 2018 Sep;13(9):2031-2061. doi: 10.1038/s41596-018-0030-9. PMID 30190556
- [Background] van den Brand R, Heutschi J, Barraud Q, DiGiovanna J, Bartholdi K, Huerlimann M, Friedli L, Vollenweider I, Moraud EM, Duis S, Dominici N, Micera S, Musienko P, Courtine G. Restoring voluntary control of locomotion after paralyzing spinal cord injury. Science. 2012 Jun 1;336(6085):1182-5. doi: 10.1126/science.1217416. PMID 22654062
- [Background] Hofstoetter US, Perret I, Bayart A, Lackner P, Binder H, Freundl B, Minassian K. Spinal motor mapping by epidural stimulation of lumbosacral posterior roots in humans. iScience. 2020 Dec 11;24(1):101930. doi: 10.1016/j.isci.2020.101930. eCollection 2021 Jan 22. PMID 33409476
- [Background] Nishioka K, Nakajima M. Beneficial Therapeutic Effects of Spinal Cord Stimulation in Advanced Cases of Parkinson's Disease With Intractable Chronic Pain: A Case Series. Neuromodulation. 2015 Dec;18(8):751-3. doi: 10.1111/ner.12315. Epub 2015 Jun 5. PMID 26047363
- [Background] Nicolelis MA, Fuentes R, Petersson P, Thevathasan W, Brown P. Spinal cord stimulation failed to relieve akinesia or restore locomotion in Parkinson disease. Neurology. 2010 Oct 19;75(16):1484; author reply 1484-5. doi: 10.1212/WNL.0b013e3181f46f10. No abstract available. PMID 20956795
- [Background] Pinto de Souza C, Hamani C, Oliveira Souza C, Lopez Contreras WO, Dos Santos Ghilardi MG, Cury RG, Reis Barbosa E, Jacobsen Teixeira M, Talamoni Fonoff E. Spinal cord stimulation improves gait in patients with Parkinson's disease previously treated with deep brain stimulation. Mov Disord. 2017 Feb;32(2):278-282. doi: 10.1002/mds.26850. Epub 2016 Nov 10. PMID 27862267
- [Background] Prasad S, Aguirre-Padilla DH, Poon YY, Kalsi-Ryan S, Lozano AM, Fasano A. Spinal Cord Stimulation for Very Advanced Parkinson's Disease: A 1-Year Prospective Trial. Mov Disord. 2020 Jun;35(6):1082-1083. doi: 10.1002/mds.28065. Epub 2020 Apr 20. No abstract available. PMID 32311155
- [Background] Maetzler W, Nieuwhof F, Hasmann SE, Bloem BR. Emerging therapies for gait disability and balance impairment: promises and pitfalls. Mov Disord. 2013 Sep 15;28(11):1576-86. doi: 10.1002/mds.25682. PMID 24132846
- [Background] Milekovic T, Moraud EM, Macellari N, Moerman C, Raschella F, Sun S, Perich MG, Varescon C, Demesmaeker R, Bruel A, Bole-Feysot LN, Schiavone G, Pirondini E, YunLong C, Hao L, Galvez A, Hernandez-Charpak SD, Dumont G, Ravier J, Le Goff-Mignardot CG, Mignardot JB, Carparelli G, Harte C, Hankov N, Aureli V, Watrin A, Lambert H, Borton D, Laurens J, Vollenweider I, Borgognon S, Bourre F, Goillandeau M, Ko WKD, Petit L, Li Q, Buschman R, Buse N, Yaroshinsky M, Ledoux JB, Becce F, Jimenez MC, Bally JF, Denison T, Guehl D, Ijspeert A, Capogrosso M, Squair JW, Asboth L, Starr PA, Wang DD, Lacour SP, Micera S, Qin C, Bloch J, Bezard E, Courtine G. A spinal cord neuroprosthesis for locomotor deficits due to Parkinson's disease. Nat Med. 2023 Nov;29(11):2854-2865. doi: 10.1038/s41591-023-02584-1. Epub 2023 Nov 6. PMID 37932548